CLINICAL TRIAL: NCT02543450
Title: Two Different Physiotherapy Programs in Order to Improve Walking Capacity and Participation in Chronic Stroke Subjects
Brief Title: Physiotherapy in Order to Improve Walking Capacity and Participation in Chronic Stroke Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Nueva Opción Brain Damage Association (Unknown)
Responsible Party: Principal Investigator, M Luz Sanchez, Profesor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stroke_Project_15
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: Chronic stroke; Participation; Walking ability
MeSH Terms: conditions — Stroke | interventions — Blood Circulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiovascular/task-oriented training (Experimental): 8 cardiovascular exercises at moderate intensity, interrupted by 1-minute active breaks of task-oriented exercises.
  Interventions: Other: Cardiovascular and task-oriented training
- Upper limb strength training program (Active Comparator): Nine 5-minute station circuit session. Patients work 2+2 minutes in each exercise, with a 30-second rest between the 2-minute periods and between stations.
  Interventions: Other: Upper limb strength training program

INTERVENTIONS:
Other: Cardiovascular and task-oriented training
  Arms: Cardiovascular/task-oriented training
Other: Upper limb strength training program
  Arms: Upper limb strength training program

SUMMARY:
In hemiplegic stroke patients, gait performance is affected by impaired walking endurance. Evidence has shown that higher exercise intensity improves cardiovascular fitness, while greater dose in task repetition benefits locomotor function. Therefore, the goal of this study is to examine the effect of a combined cardiovascular/task-oriented interval training programme on the walking capacity of chronic stroke individuals and the improvement in their participation.

DETAILED DESCRIPTION:
Owing to the high prevalence of disability in stroke older adults, walking capacity and participation can be severely affected. According to the International Classification of Functioning, Disability and Health 2001, participation involves functioning in life. In Rehabilitation Medicine, there has been a growing concern about it as a way to assess success of treatment. However, appraisal of participation in stroke research is scarce.

In all stages after a stroke, Physiotherapy interventions in favor of intensive high repetitive task-oriented and task-specific training have obtained benefits on trained actions and activities. But, the effect of this type of treatment on the impact the disease has on patient´s participation is under investigated.

The aim of this study was to determine which kind of physiotherapy task-oriented training program could better improve participation in chronic stroke subjects: an upper limb strength training program (ULST) or a combined cardiovascular/task-oriented interval training (IT) program.

Therefore, the goal of this study is to examine the effect of a combined cardiovascular/task-oriented interval training programme on the walking capacity of chronic stroke individuals and the improvement in their participation.

A randomized single-blind controlled trial was carried out. Fourteen subjects with chronic hemiplegia resulting from stroke (onset >6m) were recruited. All participants were fully informed about the experimental procedures and the aim of the study. Written informed consent was signed by each subject prior to participate. Approval from the ethics committee of the University of Valencia was obtained for the study.

Subjects were randomly allocated to an ULST program with elastic bands (n=7) or to a cardiovascular/task-oriented IT program (n=7), focused on walking capacity. In the ULST group, a nine 5-minute station circuit session was designed. Patients work 2+2 minutes in each exercise, with a 30-second rest between the 2-minute periods and between stations. The IT program consisted of a set of 8 cardiovascular exercises at moderate intensity, interrupted by 1-minute active breaks of task-oriented exercises. Duration of both programmes was 3 months (3 sessions/week).

Participation was assessed by the Stroke Impact Scale (SIS-16) and the Frenchay Activities Index (FAI), before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* More than 6 months after first stroke

Exclusion Criteria:

* Functional disability not related to the aftermath of stroke
* Participate in other rehabilitation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Participation (Frenchay Activities Index (FAI)) | At 3 months
  Frenchay Activities Index (FAI)

SECONDARY OUTCOMES:
Walking ability | At 3 months
  6 min-walk
Upper limb function (Fugl-Meyer Assessment) | At 3 months
  Fugl-Meyer Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Sánchez-Sánchez ML, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

REFERENCES:
- [Derived] Sanchez-Sanchez ML, Ruescas-Nicolau MA, Perez-Miralles JA, Marques-Sule E, Espi-Lopez GV. Pilot randomized controlled trial to assess a physical therapy program on upper extremity function to counteract inactivity in chronic stroke. Top Stroke Rehabil. 2017 Apr;24(3):183-193. doi: 10.1080/10749357.2016.1245395. Epub 2016 Oct 19. PMID 27760505